CLINICAL TRIAL: NCT07048990
Title: The Effects of Empowerment Group Therapy on Ukrainian Adult Outpatients Located Inside the Country During the War
Brief Title: Feasibility of Empowerment Group Therapy on Ukrainian Adult Outpatients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Solveig Kemna, Resident/research associate, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMPOWER_UA_ADULTS_2025
Record Dates: First submitted 2025-06-18; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Depression NOS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-based group therapy intervention "Empowerment" (Experimental): 10 CBT-based psychotherapeutic group sessions will be held weekly, either in person or online, through trained psychiatrists or psychotherapists from the Department of Medical Psychology, Psychosomatic Medicine, and Psychotherapy at Bogomolets National Medical University.
  During the first group session, participants will receive the workbook "Empowerment" ("Опора та стійкість"), which is to be completed at home between sessions as homework. Each session will include an assessment of the participants' general current condition, their engagement in the psychotherapeutic interventions, group dynamics, and more.
  Interventions: Behavioral: Empowerment Group Therapy

INTERVENTIONS:
Behavioral: Empowerment Group Therapy — Empowerment is a manualized, culturally sensitive treatment program. The treatment is based on a modular principle that transdiagnostically targets major symptom domains (e.g. stress, depression, anxiety), and can be flexibly adapted to individual mental health conditions of clients who participate in this program. The intervention is designed as a psychological group intervention for resource-limited settings and scalable for different formats (i.e. in-person, online, hybrid) to be feasible under the unstable conditions of war (e.g. missile attacks, power outrages). Key therapeutic elements are psychoeducation, emotion regulation strategies, problem solving and building coping skills. The activation of individual and culture-specific resources as well as building self-help skills are at focus of the treatment.

SUMMARY:
This single-arm pilot study aims to explore the feasibility and acceptability of the culturally adapted, Ukrainian version of the Empowerment Group Therapy (Wiechers, 2023) manual and accompanying workbook for the Ukrainian population affected by the ongoing war. Feasibility will be evaluated based on participant retention. Acceptability will be assessed through questionnaires and qualitative feedback. The study also gathers preliminary data on the effectiveness of the intervention by assessing changes in quality of life, stress, symptoms of anxiety, depression, PTSD, and somatization. Overall, it seeks to explore the relevance and impact of group-based resilience therapy in a conflict-affected setting.

DETAILED DESCRIPTION:
The investigators will identify eligible participants at the Bogomolets outpatient department. An eligibility screening conducted in person to ensure the inclusion criteria are met. All participants must sign an informed consent form after receiving written and verbal study information. Participants will carry out self-reported measurements at baseline (T0), after the intervention phase of 10-11 weeks (T1), and at follow-up at 4 weeks after the last intervention session (T2). The participants receive ten group therapy sessions, which are delivered in an in-person or digital setting. The intervention will be provided for five groups, each comprised of 10 to 14 participants, including overall 50 to 70 persons.

The Empowerment intervention (Wiechers 2023) is a depression-specific CBT-based group therapy. It is based on 16 modules which can be selected according to the needs of the group. The sessions start with a mindfulness or breathing exercise, and focus on psychoeducation and behavioral activation. The manual was culturally adapted to the current Ukrainian context and translated into Ukrainian.

The data management plan includes standard procedures for data-handling such as using anonymized identification codes for patient data. Besides, the participants have the right to access their data, and the right to claim an annihilation. The data is being saved in an online database, only allowing researchers involved in the study to access the data.

ELIGIBILITY:
Inclusion Criteria:

* Civilians
* 18 years of age or older
* Residency in Ukraine at the onset of the full-scale war in Ukraine and at the time of the study
* Ability to participate in in-person or online sessions
* Ability to participate in online sessions, including communication via smartphone chat
* Speaks Ukrainian or Russian
* Presence of depression, anxiety, stress according to DSM-5 criteria, or psychological distress directly or indirectly caused by the war (other conditions may be included if deemed appropriate by a physician)
* Moderate severity of symptoms on the depression, anxiety, or stress subscale of the DASS-21
* Anyone who, upon being placed on the waiting list, recognizes a need for help and support is eligible to participate
* Signed informed consent form

Exclusion Criteria:

* Lack of informed consent
* Diagnosis of schizophrenia, autism spectrum disorders, degenerative disorders, or significant cognitive impairments
* Use of psychoactive substances and alcohol
* Acute risk of suicide
* Ongoing psychotherapy or psychotherapy within the past 3 months
* Psychopharmacological treatment (at the discretion of the therapist during screening)
* Current inpatient treatment
* Incomplete screening questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Post-Intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline)
  Feasibility will be indexed by inclusion rate of participants to the study.
Feasibility of the intervention | Post-Intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline)
  Feasibility will be indexed by participants attendance of the group therapy sessions (>80% of sessions).
Feasibility of the intervention | Post-Intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline)
  Feasibility will be indexed by droup-out rate (<20% of participants).
Acceptability of the intervention | Post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline)
  Acceptability will be assessed by the rate of intervention completion (>80% complete all sessions).
Acceptability of the intervention | Post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline)
  Acceptability will be assessed by using the Client Satisfaction Questionnaire (Attkisson & Zwick, 1982).

SECONDARY OUTCOMES:
Stress, anxiety and depression | At baseline, post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline), and follow-up (4 weeks after last group therapy session)
  The Depression Anxiety Stress Scale (Nilges & Essau, 2015) will be used to analyse symptoms of stress, anxiety and depression. The score ranges from 0 to 63, with higher scores indicating higher levels of depressive and anxiety symptoms.
Depressive symptoms | At baseline, post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline), and follow-up (4 weeks after last group therapy session)
  The Patient Health Questionnaire - 9 (Kroenke, 2001) will be used to assess depressive symptoms. Scores range from 0 to 27. Higher scores indicate greater severity of depression.
PTSD Symptoms | At baseline, post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline), and follow-up (4 weeks after last group therapy session)
  The Posttraumatic Stress Disorder Checklist for DSM-5 (Blevins, 2015) will be used to analyse symptoms of PTSD. The symptom severity score ranges from 0 to 80 with higher scores indicating higher symptom levels.
Somatic symptom burden | At baseline, post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline), and follow-up (4 weeks after last group therapy session)
  The Somatic Symptom Scale-8 (Gierk 2013) will be used to assess somatic symptom burden. Scores range from 0 to 32, with higher scores indicating greater somatic symptom burden
Health-related Quality of Life | At baseline, post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline), and follow-up (4 weeks after last group therapy session)
  The 36-Item Short Form Health Survey (Ware & Sherbourne 1992) will be used to assess health-related quality of life. Each of the eight health domains in the SF-36 is scored on a 0 to 100 scale, where 0 represents the worst possible health status and 100 represents the best possible health status.
Resilience | At baseline, post-intervention (after completion of 10 group psychotherapy sessions; 10 to 11 weeks from baseline), and follow-up (4 weeks after last group therapy session)
  The Brief Resilience Scale (Smith 2009) will be used to assess the ability to bounce back or recover from stress. The scale consists of six items rated on a 5-point Likert scale. For interpretation, a mean score is calculated ranging from 1 to 5, with higher scores indicating greater resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical University Bogomolets, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided